CLINICAL TRIAL: NCT00823693
Title: Multi-center, Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Safety and Efficacy of Bimosiamose 5% Cream for the Treatment of Patients With Chronic Plaque Type Psoriasis
Brief Title: Safety and Efficacy Study of Bimosiamose Cream to Treat Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revotar Biopharmaceuticals AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R013
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bimosiamose Cream (Active Comparator)
  Interventions: Drug: Bimosiamose Cream
- Placebo Cream (Placebo Comparator)
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: Bimosiamose Cream
  Arms: Bimosiamose Cream
Drug: Placebo Cream
  Arms: Placebo Cream

SUMMARY:
The purpose of this study is to determine whether Bimosiamose Cream is safe and effective in the treatment of plaque type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque type psoriasis PASI score of 5-15
* At least 18 years of age
* Written informed consent

Exclusion Criteria:

* Active skin infection
* More than 20% Body Surface Area (BSA) affected by psoriasis
* Use of certain anti-psoriasis medication or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Mitte, Klinik für Dermatologie, Venerologie und Allergologie, Berlin, Germany